CLINICAL TRIAL: NCT04150809
Title: A Non-Interventional Pilot Study to Explore the Role of Gut Flora in Amyotrophic Lateral Sclerosis
Brief Title: A Study to Explore the Role of Gut Flora in ALS
Status: Withdrawn | Type: Observational
Why Stopped: Company shifted focus
Sponsor: ProgenaBiome (Other)
Responsible Party: Sponsor
Other Study IDs: PRG-024
Record Dates: First submitted 2019-10-30; First posted 2019-11-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: ALS; Amyotrophic Lateral Sclerosis; Motor Neuron Disease
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool Samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: Patients who have been diagnosed with ALS.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — There is no intervention for this study

SUMMARY:
This study seeks to correlate microbiome sequencing data with information provided by patients and their medical records regarding ALS

DETAILED DESCRIPTION:
The goal of this Research Study is to better understand how the genetic information in subject's microbiome correlates to the information provided in surveys and in medical records regarding ALS

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent, demonstrating that the patient understands the procedures required for the study and the purpose of the study
2. Male or female patients of any age (interest is given to children to compare with mothers).
3. Diagnosis of ALS

Exclusion Criteria:

1. Refusal to sign informed consent form
2. History of bariatric surgery, total colectomy with ileorectal anastomosis or proctocolectomy.
3. Postoperative stoma, ostomy, or ileoanal pouch
4. Participation in any experimental drug protocol within the past 12 weeks
5. Treatment with total parenteral nutrition
6. Any clinically significant evidence of disease that could interfere with the subject's ability to enter the trial
7. Inability to adequately communicate with the investigator or their respective designee and/or comply with the requirements of the entire study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with ALS
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2030-03 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Correlation of Microbiome to ALS via Relative Abundance Found in Microbiome Sequencing | One year
  The identification of bacterial species residing the gut flora will be processed by next generation sequencing followed by metagenomic analysis. Bacterial diversity will then be evaluated in parallel with relative abundance of targeted species within and among individual microbes. In other words, in patients with ALS a specific microbe or class of microbes might represent a larger percentage of the microbiome when compared to healthy individuals. There could also be a higher or lower Shannon Index.

SECONDARY OUTCOMES:
Validation of Sequencing Methods | One year
  To validate the methods used to sequence sample

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Hazan, MD, Principal Investigator — ProgenaBiome
Locations (1):
- ProgenaBiome, Ventura, California, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD